CLINICAL TRIAL: NCT06122883
Title: Official Title Evaluating the Effect of Dentist's Attire on Children's Acceptance of Dental Treatment Including Local Anesthesia
Brief Title: Dental Attire Effect on Children's Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Pedo-10-2023
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Behavior, Child; Dental Anxiety; Anesthesia, Local
Keywords: Dental attire; Behavior management; Children fear
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Distraction in the reception area. (Experimental)
  Interventions: Behavioral: Evaluation the effectiveness of distraction in the reception area in the management of anxious pediatric patients during dental local anesthesia
- Distraction in the treatment area. (Experimental)
  Interventions: Behavioral: Evaluation the effectiveness of distraction in the treatment area in the management of anxious pediatric patients during dental local anesthesia
- Distraction in both treatment and reception area. (Experimental)
  Interventions: Behavioral: Evaluation the effectiveness of distraction in both reception and treatment areas in the management of anxious pediatric patients during dental local anesthesia
- Basic behavior guidance techniques without using any type of distraction aids. (Other)
  Interventions: Behavioral: Evaluation of the effectiveness of basic behavior guidance techniques without using any type of distraction aids in the management of anxious pediatric patients during dental local anesthesia

INTERVENTIONS:
Behavioral: Evaluation the effectiveness of distraction in the reception area in the management of anxious pediatric patients during dental local anesthesia — Buccal and palatal infiltration will be administrated with basic behavior guidance techniques while the dentist wearing conventional attire in the treatment room after meeting the child in the reception area while wearing the friendly attire.
  Arms: Distraction in the reception area.
Behavioral: Evaluation the effectiveness of distraction in the treatment area in the management of anxious pediatric patients during dental local anesthesia — Buccal and palatal infiltration will be administrated with basic behavior guidance techniques while the dentist wearing friendly attire in the treatment room after meeting the child in the reception area while wearing the conventional attire.
  Arms: Distraction in the treatment area.
Behavioral: Evaluation the effectiveness of distraction in both reception and treatment areas in the management of anxious pediatric patients during dental local anesthesia — Buccal and palatal infiltration will be administrated with basic behavior guidance techniques while the dentist wearing friendly attire in the reception area and treatment room.
  Arms: Distraction in both treatment and reception area.
Behavioral: Evaluation of the effectiveness of basic behavior guidance techniques without using any type of distraction aids in the management of anxious pediatric patients during dental local anesthesia — Buccal and palatal infiltration will be administrated with basic behavior guidance techniques while the dentist wearing conventional attire in the reception area and treatment room.
  Arms: Basic behavior guidance techniques without using any type of distraction aids.

SUMMARY:
The aim of this study is to evaluate the effect of friendly attire on dental anxiety among children visiting dental office in comparison with conventional attire. All of the children who will be experienced maxillary dental anesthesia with/without distraction will be assessed by using a combination of measures: Wong-Baker faces and the Children's Fear Scale (self-report), heart pulse rate, and behavior (using Anxiety levels using Face - Legs - Activity - Cry - Consolability "FLACC" scale "external evaluator") Acceptance will be measured using a two-point Likert scale.

DETAILED DESCRIPTION:
This study will evaluate the effect of dental attire on children's acceptance of different dental treatments that include dental anesthesia. pain and anxiety will be evaluated during buccal and palatal infiltration using five behavioral scales, Wong-Baker pain scale, Children's Fear Scale and Children's Anxiety Questionnaire (self-report), pulse rate (physiological) and behavior (using FLACC behavior rating scale "external evaluator".

Heart pulse rate measurement will be recorded firstly when the patient is seated comfortably in the reception area, on dental chair prior to the injection, and finally after the procedure is done and the child patients will be asked to choose a face that describe their status from one of both Wong Baker faces scale, Children's Fear Scale and Children's Anxiety Questionnaire.

Body responses of all child patients will be recorded during the whole procedure and then will be evaluated by an external evaluator to determine the children behavioral score according to FLACC scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 and 10 years.
2. No previous dental experience.
3. Definitely positive or positive according to Frank scale.
4. Need of maxillary anesthesia for any dental treatment.

Exclusion Criteria:

1. Previous dental experience
2. Systematic or mental disorders.
3. Definitely negative or negative according to Frankel scale

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Pain levels | 5 minutes following the dental local anesthesia.
  Pain levels will be measured by using a self-reported simplified Wong-Baker faces pain scale:
  0 no Hurt - 1 Hurts little Bit - 2 Hurts little More - 3 Hurts Even More - 4 Hurts Whole Lot - 5 Hurts Worst
Anxiety levels | 1 minute during the dental local anesthesia.
  This will be evaluated using the Face-Legs-Activity-Cry-Consolability (FLACC) scale (0 low anxiety and pain level - 10 high anxiety and pain level).
Anxiety levels | 5 minutes following the meeting with the dentist in the reception area, and 5 minutes after the patient is seated comfortably on the dental chair
  This will be evaluated using Children's Fear Scale (0 indicating 'no anxiety' and 4 indicating 'extreme anxiety') and Children Anxiety Questionnaire (self-report) (4 indicating 'no anxiety' and 16 indicating 'extreme anxiety').
Pulse rate | (1) five minutes after the patient is seated comfortably in the reception area, (2) five minutes after the patient is seated comfortably on the dental chair, (3) five minutes following the injection of the anesthetic drug
  Pulse rate (the number of times your heart beats each minute bpm will be evaluated using Finger Pulse Oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Jamila Bchara, DDs, Principal Investigator — Damascus University; Mohannad Laflof, Phd, Study Director — Damascus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kastelic DR, Volpato LE, de Campos Neves AT, Aranha AM, Martins CC. Do Children and Adolescents Prefer Pediatric Attire over White Attire during Dental Appointments? A Meta-analysis of Prevalence Data. Int J Clin Pediatr Dent. 2021 Jan-Feb;14(1):14-29. doi: 10.5005/jp-journals-10005-1861. PMID 34326579
- [Background] Kamavaram Ellore VP, Mohammed M, Taranath M, Ramagoni NK, Kumar V, Gunjalli G. Children and Parent's Attitude and Preferences of Dentist's Attire in Pediatric Dental Practice. Int J Clin Pediatr Dent. 2015 May-Aug;8(2):102-7. doi: 10.5005/jp-journals-10005-1293. Epub 2015 Aug 11. PMID 26379376
- [Background] Festini F, Occhipinti V, Cocco M, Biermann K, Neri S, Giannini C, Galici V, de Martino M, Caprilli S. Use of non-conventional nurses' attire in a paediatric hospital: a quasi-experimental study. J Clin Nurs. 2009 Apr;18(7):1018-26. doi: 10.1111/j.1365-2702.2008.02430.x. PMID 19284436
- [Background] Babaji P, Chauhan PP, Rathod V, Mhatre S, Paul U, Guram G. Evaluation of child preference for dentist attire and usage of camouflage syringe in reduction of anxiety. Eur J Dent. 2017 Oct-Dec;11(4):531-536. doi: 10.4103/ejd.ejd_223_17. PMID 29279683
- [Background] Dionigi A, Sangiorgi D, Flangini R. Clown intervention to reduce preoperative anxiety in children and parents: a randomized controlled trial. J Health Psychol. 2014 Mar;19(3):369-80. doi: 10.1177/1359105312471567. Epub 2013 Jan 29. PMID 23362335
- [Background] Manyande A, Cyna AM, Yip P, Chooi C, Middleton P. Non-pharmacological interventions for assisting the induction of anaesthesia in children. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD006447. doi: 10.1002/14651858.CD006447.pub3. PMID 26171895